CLINICAL TRIAL: NCT07047404
Title: A Multicentre, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of BP1.4979 in Adult Patients With Primary Premature Ejaculation
Brief Title: Proof of Concept Study on BP1.4979 Effect on Primary Premature Ejaculation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P24-04/BP1.4979
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Premature (Early) Ejaculation
Keywords: premature (early) ejaculation; primary premature ejaculation; Lifelong premature ejaculation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Multicentre, randomized, double-blind, placebo-controlled, parallel-group, proof of concept study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BP1.4979 (Experimental): One tablet of BP1.4979 taken per requested need about 2 hours prior to sexual intercourse and at a 12-hour interval minimum over 12 weeks
  Interventions: Drug: BP1.4979
- Placebo (Placebo Comparator): One tablet of matching placebo taken per requested need about 2 hours prior to sexual intercourse and at a 12-hour interval minimum over 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BP1.4979 — selective dopamine D3 partial agonist
  Arms: BP1.4979
Drug: Placebo — matching placebo of BP1.4979 30mg tablet
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if drug BP1.4979 works to treat primary premature ejaculation in adults. It will also learn about the safety of drug BP1.4979. The main questions it aims to answer are:

* Does drug BP1.4979 increase the time to ejaculation during sexual intercourse?
* Do participants have a good safety and tolerability of drug BP1.4979? Researchers will compare drug BP1.4979 to a placebo (a look-alike substance that contains no drug) to see if drug BP1.4979 works to treat primary premature ejaculation.

Participants will:

* Take drug primary premature ejaculation or a placebo per requested need prior to sexual intercourses for 12 weeks
* Visit the clinic 4 times for checkups and questionnaires completion and have 2 phone calls with the study team over a period of about 17 weeks
* Keep a diary of the intakes of the experimental drug, ejaculation time, ejaculation control, any unusual events concerning their health and any other medication taken

DETAILED DESCRIPTION:
Premature ejaculation is meant when ejaculation occurs too quickly during sexual activity with a partner, often within one minute of penetration, in 75-100% of sexual encounters and for no other reason. This can be a source of frustration and distress for both partners. There are two main types of PE: lifelong (primary) PE, present from the first sexual experience, and acquired (secondary) PE, which develops later in life and is often associated with other sexual problems (such as reduced libido or erectile dysfunction).

The exact cause of PE remains poorly understood. In the case of primary PE, it may be linked to brain chemicals (such as serotonin and dopamine), nervous system problems or psychological factors.

Current treatments include drugs and non-drug therapies. Medication works by increasing serotonin levels in the brain. They may be authorised, such as dapoxetine (a short-acting antidepressant) and anaesthetic creams (often used to reduce sensitivity, e.g. prilocaine-lidocaine), or prescribed off-label, such as other antidepressants or analgesics (e.g. tramadol). However, these treatments are often of limited efficacy, leaving patients without satisfactory solution.

The objective of this trial is to develop an effective treatment for primary PE specifically and to address an unmet medical need by improving the quality of life of the patients concerned.

The drug under study, called BP1.4979, acts on the dopamine pathway and is being tested to assess whether it can help men suffering from primary PE to better control their ejaculation. The study will compare BP1.4979 with a placebo (a tablet that looks identical but has no active ingredient), taken on demand before sexual intercourse, over a 12-week period.

The study is a double-blind trial compared to a placebo, which means that neither the participants nor the study doctors know who is receiving the study drug or the placebo so as not to influence the results obtained. The treatments will be assigned randomly (by drawing lots), thus forming one group receiving BP1.4979 and another receiving the corresponding placebo.

A visit to the clinical site is planned at the beginning of the selection phase. Participants will be asked to sign an informed consent form prior to any study-related procedure. During the screening phase, they will use a stopwatch to measure the time to ejaculation during sex with a female partner over a period of approximately four weeks and record these times in a diary.

Patients will then return to the clinical site to check whether they are eligible to take part in the study at the 'randomisation visit' and, if so, they will receive the study drug for one month's treatment.

Follow-up visits will take place at week 4 (safety tests and renewal of treatment for two months) and week 12 (final visit). A telephone call will be made at week 8 and week 13 (7 days after stopping treatment) to check or monitor any side effects.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18 to 50 years old (both inclusive)
* Diagnosis of primary (lifelong) PE according to the investigator
* Intravaginal Ejaculatory Latency Time (IELT) estimated by the patient around one (1) minute at screening
* Confirmation at randomization visit that at least 3 timed sexual intercourses with each IELT below 90 seconds occurred during the baseline period
* Patient must be able to provide an informed consent and voluntarily express a willingness to participate in this study, and must sign and date an informed consent prior to any study specific procedure
* Capability to participate in all study tests according to the investigator

Exclusion Criteria:

* Diagnosis of acquired PE, pseudo-PE or natural variable PE
* History of clinically significant abnormalities comprising cardiovascular (including especially prolonged QTc (>450 ms) and high degree (second and third) atrio-ventricular blocks)), hematological, neurological, and endocrine diseases
* Current therapy with any treatment which may impact PE from 4 weeks prior to the screening visit
* Current therapy with any treatment displaying dopamine D3 receptor agonist properties from 4 weeks prior to the screening visit
* Concomitant intake of psychoactive / chem-sex substances

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Intravaginal ejaculatory latence time (IELT) | 12 weeks
  IELT measured with a stopwatch started by the partner at vaginal intromission and stopped at the start of intravaginal ejaculation at each sexual encounter

OTHER OUTCOMES:
Ejaculatory control score per sexual encounter | 12 weeks
  For each sexual encounter, with or without IMP intake, the patient will grade and report in the diary a 4-point ejaculatory control Likert scale, stated as follows "During this sexual intercourse, was your control over ejaculation: 1-Very poor, 2-Poor, 3-Good, 4-Very good or "No opinion"
Ejaculatory control | At randomization, visit 2 (4 weeks) and end of treatment visit (12 weeks)
  5-point ejaculatory Likert scale evaluating the overall impact of the IMP during the previous month.
  The question is worded as follows: "Did you have a lack of ejaculatory control or ability to postpone ejaculation during the last month?", the answers being: 0: Almost all of the time (>80%), 1: Most of the time (60-80%), 2: About half of the time (40-60%), 3: Less than half of the time (20-40%), 4: Close to never (<20%)". Higher scores thus indicate a lower frequency of premature ejaculation.
Male Sexual Health Questionnaire | At randomization visit, visit 2 (at 4 weeks) and end of treatment visit (at 12 weeks)
  25-item self-administered questionnaire aiming at assessing erection, ejaculation, satisfaction and sexual activity and desire over the previous month
Patient Global Impression Scale - Improvement (PGI-I) | Visit 1 (Randomization), Visit 2 (4 weeks) and end of treatment visit (12 weeks)
  one item adapted to the patient, to assess if there's been an improvement in his clinical status since the IMP intake.
  The patient will be asked at Visit 2 and EoT (Visit 4) to select the number that best describes how he has felt during the previous month in comparison to the study onset: 0 = Not assessed, 1 = Very much better, 2 = Much better, 3 = A little better, 4 = The same, 5 = A little worse, 6 = Much worse, 7 = Very much worse.
Safety assessed by Adverse Event (AEs) collection | 12 weeks
  Safety of BP1.4979 based on AEs reporting during the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Study principal investigator, Principal Investigator — University hospital of Nîmes
Locations (1):
- University Hospital of Nîmes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No